CLINICAL TRIAL: NCT03309800
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled, Parallel, Phase II Clinical Trial to Evaluate the Efficacy and Safety of HL301 Versus Placebo in Acute Bronchitis Patients
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of HL301 Versus Placebo in Acute Bronchitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL_HL301_202
Record Dates: First submitted 2017-09-08; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Acute Bronchitis
Keywords: Acute Bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): HL301: 2Tab/day: 1 Tablet at once, 2 times a day, 7 days of treatment
  Interventions: Drug: HL301
- Placebo comparator (Placebo Comparator): HL301(Placebo): 2Tab/day: 1 Tablet at once, 2 times a day, 7 days of treatment
  Interventions: Drug: HL301(Placebo)

INTERVENTIONS:
Drug: HL301 — HL301: 2Tab/day: 1 Tablet at once, 2 times a day, 7 days of treatment
  Arms: Experimental
Drug: HL301(Placebo) — HL301(Placebo): 2Tab/day: 1 Tablet at once, 2 times a day, 7 days of treatment
  Arms: Placebo comparator

SUMMARY:
A Multicenter, Randomized, Double-blinded, Placebo-controlled, Parallel, Phase II Clinical Trial to Evaluate the Efficacy and Safety of HL301 versus Placebo in acute bronchitis patients.

Endpoint: BSS, The improvement and improvement rate of the tester for the treatment response, The satisfaction of the subject, Total usage of Acetaminophen

ELIGIBILITY:
Inclusion Criteria:

1. Both gender, 19 years ≤ age ≤ 80 years
2. (Bronchitis Severity Score)* ≥ 5point at Visit 2 (Randomized Visit)
3. Acute bronchitis within 48hr based on Visit 2 (Randomized Visit)
4. Those who can comply with the requirements of clinical trials
5. Written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

1. Patients with respiratory and systemic infections requiring systemic antibiotic therapy
2. Patients with bleeding tendency
3. Patients who investigators determines to severe respiratory disease that would interfere with study assessment
4. Patients who were treated with oral systemic adrenocortical hormone or immunosuppressive drug within 4 weeks prior to Visit 2
5. Patients who were treated with oral antihistamines, ACE suppressive. or systemic/inhalative glucocorticosteroid within 2 weeks prior to Visit 2

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Bronchitis Severity Total Score(BSS) Change | Visit 1 (-3 day), Visit 2 (0 day), Visit 3 (7 day)
  Evaluation period: Visit 1 (-3 day), Visit 2 (0 day), Visit 3 (7 day)

SECONDARY OUTCOMES:
The improvement and improvement rate of the tester for the treatment response (Chi-square test or Fisher's Exact test) | Visit 3 (7 day)
  Evaluation period: Visit 3 (7 day)
The satisfaction of the subject (Questionnaire) | Visit 3 (7 day)
  Evaluation period: Visit 3 (7 day)
Total usage of Acetaminophen | Visit 3 (7 day)
  Evaluation period: Visit 3 (7 day)

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital, Seoul, Dongdaemun-gu, South Korea